CLINICAL TRIAL: NCT07072650
Title: Impact of Adding Dexmedetomidine as an Adjuvant to The Local Anesthetic in QL3 in Patient Undergoing Caesarean Section
Brief Title: Impact of Adding Dexmedetomidine as an Adjuvant to The Local Anesthetic in Quadratus Lumborum Block in Patient Undergoing Caesarean Section
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Majid Fakhir Mutar Alhamaaidah (Other)
Responsible Party: Sponsor-Investigator, Majid Fakhir Mutar Alhamaaidah, Head of Scientific committee, Dep. of Anesthesiology, Principal Investigator, Al-Ayen Iraqi University
Organization: Al-Ayen Iraqi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4/2025 in 7/01/2025
Record Dates: First submitted 2025-06-28; First posted 2025-07-18 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-07

CONDITIONS: Dexmedetomidine; Quadratus Lumborum Block; Postoperative Analgesia; Caesarean Section
Keywords: dexmedetomidine; Quadratus lumborum block; caesarean section
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group dB (Active Comparator): Adding Dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- Group B (No Intervention): Only bupivacaine

INTERVENTIONS:
Drug: Dexmedetomidine — Studying combining a local anesthetic with dexmedetomidine (DEX) in a quadratus lumborum block (QLB) following a cesarean section (CS) in elective surgery in Bint Al-Huda Hospital.
  Arms: Group dB

SUMMARY:
The goal of this clinical trial is to evaluate the effects of adding Dexmedetomidine to local anesthetic agent (bupivacaine) for quadratus lumborum block (QLB) after spinal anesthesia in patient undergoing elective caesarean section. The main questions it aims to answer are:

1. does adding dexmedetomidine enhance analgesia time?
2. does adding dexmedetomidine reduce recovery time?
3. does adding dexmedetomidine lower the need of analgesic medication after surgery? Study include 80 female pregnant non-obese patients scheduled for elective caesarean section.

DETAILED DESCRIPTION:
Effective postoperative analgesia facilitates a mother's quick recovery, enhances early ambulation, promotes breastfeeding, and reduces the risk of postoperative thromboembolism. The aim of this study was to evaluate the postoperative analgesic efficacy of combining a local anesthetic with dexmedetomidine (DEX) in a quadratus lumborum block (QLB) following a cesarean section (CS). A prospective, randomized, blind, controlled trial included 80 female patients aged 18 - 40 years old who underwent cesarean delivery under spinal anesthesia, were randomly assigned to two equal groups. Group dB received a quadratus lumborum block (QLB) with 20 ml of 0.25% bupivacaine and dexmedetomidine (0.5 μg/kg) on each side, while Group B received QLB with 20 ml of 0.25% bupivacaine alone on each side. The primary outcome measured was total analgesic consumption over 24 hours postoperatively. Secondary outcomes included Visual Analog Scale (VAS) scores, time to first analgesic request, and the incidence of side effects such as sedation, nausea, vomiting, shivering, pruritus, bradycardia, hypotension, and respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years' old and less 40 years.
* With body mass indices (BMI) between 18.5 and 34.9 kg/m²
* Pregnancy more than 37 weeks with single fetus.
* Intact membranes.
* Women with a singleton pregnancy.

Exclusion Criteria:

* ASA class III or higher,
* contraindications to spinal anesthesia,
* mental or neurological disorders,
* chronic heart, renal, or liver diseases,
* emergency surgery,
* a history of blood coagulation disorders,
* allergies or contraindications to the study drugs,

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
The primary outcome measured was the postoperative pain level score. The Visual Analog Scale (VAS) was used for assessment, where 0 represented no pain and 10 represented the worst pain. | The first 24 hours postoperatively

SECONDARY OUTCOMES:
The time to the first analgesic request (within the first 24 hours postoperatively ) | over the first 24 hours postoperatively
The total analgesic consumption | Over the first 24 hours postoperatively
Sedation levels | At 2, 4, 6, 12, and 24 hours postoperatively
  Sedation levels were also monitored using the Ramsay Sedation Scale which helps assess the patient's level of sedation and consciousness; was used to assess postoperative sedation at 2, 4, 6, 12, and 24 hours postoperatively
Postoperative nausea and vomiting (PONV) | Within the first 24 hours
Mean Blood Pressure (MBP) | Perioperative period at intervals of 0, 5, 10, 20, and 30 minutes
  Measured in mmHg
Heart Rate (HR) | Perioperative period at intervals of 0, 5, 10, 20, and 30 minutes
  Measured as beats/minute

CONTACTS AND LOCATIONS:
Locations (1):
- Bint Al-Huda Hospital/ thi qar office directorate, Nasiriyah, Thi Qar, Iraq

IPD SHARING:
Plan to Share IPD: Undecided